CLINICAL TRIAL: NCT02680392
Title: Functional Outcome and Postoperative Analgesia in Total Knee Arthroplasty: a Comparison Between Continuous Adductor Canal Block and Pulsed and Thermal Radiofrequency of Saphenous and Genicular Nerves of the Knee
Brief Title: Functional Outcome and Analgesia in TKA: Radiofrequency vs Continuous Adductor Canal Block
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: McGill University Health Centre/Research Institute of the McGill University Health Centre (Other)
Responsible Party: Principal Investigator, JF Asenjo, Professor, McGill University Health Centre/Research Institute of the McGill University Health Centre
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 15-209-MUHC
Record Dates: First submitted 2016-01-19; First posted 2016-02-11 (Estimated); Last update posted 2021-10-01 (Actual); Status verified 2021-09

CONDITIONS: Osteoarthritis, Knee
Keywords: Pulsed and Continuous Radiofrequency Treatment; Continuous adductor canal block; Postoperative pain; Functional recovery; Total Knee Joint Replacement
MeSH Terms: conditions — Osteoarthritis, Knee; Pain, Postoperative | interventions — Heart Rate

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Pulsed and Continuous Radiofrequency (Experimental): In this group of patients undergoing total knee arthroplasty (allocation of patients is randomized), Pulsed radiofrequency (PRF) is applied to the saphenous nerve of the knee, associated to Continuous Radiofrequency (TRF) applied to the genicular nerves of the knee . A sham catheter is inserted in the mid-tigh to simulate a continuous adductor canal block, and connected to an infusion of normal saline (assessor and patient blinded to the treatment)
  Interventions: Procedure: Pulsed and Continuous Radiofrequency
- Continuous adductor canal block (Active Comparator): Continuous Adductor Canal Block
  Continuous adductor canal block is performed in this group of patients, with a catheter infusing ropivacaine 0.2% in the first 48 hours after surgery.
  The solutions bags are labelled in order to make assessor and patients, blinded to the treatment (Ropivacaine vs Normal Saline)
  Interventions: Drug: Continuous Adductor Canal Block

INTERVENTIONS:
Procedure: Pulsed and Continuous Radiofrequency — Preoperative pulsed radiofrequency of the saphenous nerve and Continuous radiofrequency of the genicular nerves of the knee joint.
  The saphenous nerve will be approached at the adductor canal and it will be treated with Pulsed RF for 4 minutes at 42 Celsius degrees. Ropivacaine 0.5% 10ml with Dexamethasone 10mg will be injected after the RF.
  The Genicular terminal branches of the sciatic and femoral nerves will be treated with Continuous RF for 3 min at 80 Celsius degrees and then with 2 ml of Ropivacaine 0.5% and 10 mg of Methylprednisolone to each nerve (5 in total) A sham catheter in the mid-thigh will be placed for patients in the RF group, infusing Normal Saline 0.9% and simulating a Continuous Adductor Canal Block. To blind the investigator to the type of treatment for the postoperative assessment , every solution bag will be prepared by the Pharmacy of the Hospital, covered with a plastic envelope and labeled as "Study Solution".
  Other Names: PRF
  Arms: Pulsed and Continuous Radiofrequency
Drug: Continuous Adductor Canal Block — The patients in the Adductor canal group, will have a catheter for peripheral nerve block inserted under strict asepsis in the adductor canal under ultrasound guidance, and will receive for postoperative analgesia a 48-h continuous infusion of Ropivacaine 0.2% at 8 ml/hour The patients will receive, intraoperatively 10 mg of Dexamethasone i.v.
  To blind the investigator who will do the postoperative assessment to the type of treatment, every solution bag will be prepared by the Pharmacy of the Hospital, covered with a plastic envelope and labeled as "Study Solution". It will be always possible to crack the code and find out to which group the patient belongs
  Other Names: CACB
  Arms: Continuous adductor canal block

SUMMARY:
This randomized, double blind controlled trial is designed to investigate the potential benefits of radiofrequency in terms of analgesia and functional outcome, compared to the conventional continuous adductor canal block, for patients undergoing total knee arthroplasty for osteoarthritis.

DETAILED DESCRIPTION:
The aim of this study is to compare the efficacy of two analgesia techniques in patients undergoing Total Knee Arthroplasty (TKA) on the functional recovery and pain control: Pulsed and Continuous Radiofrequency (PRF and TRF) applied respectively to the saphenous nerve and to the genicular nerves of the knee (femoral and sciatic branches) compared with Continuous adductor canal block with local anesthetics (CACB).

The Null Hypothesis is that no difference exists in the functional recovery, in pain medication consumption and in postoperative exercise and physical performance between two groups of patients submitted to TKA with the two different modalities of analgesia.

To test the null hypothesis we hypothesize as clinically relevant:

* a reduction of 30% in the time needed to perform the Timed Up and Go test at 2 days after surgery
* a reduction of 30% in pain medication consumption in the first 24 ore after surgery.

To test the null Hypothesis, 40 patients are needed (20 for each group).

The primary outcome measures will be:

* the time required in the two groups (CACB-group and RF-group) to perform the Timed-Up and Go (TUG) test on the second postoperative day (POD2). TUG measures the time that a person takes to rise from a chair, walk three meters, turn around, walk back to the chair, and sit down. During the test, the person is expected to use any mobility aids that they would normally require.
* the total morphine consumption by means of the patient-controlled analgesia pump over the first 24-h after surgery, which can be measured precisely through the record of the dose delivered by the PCA pump. With an alpha error of 0.05, a power of 80% and a standard deviation of 7 mg of morphine consumption per 24 h, 20 patients (10 in each group) will be required for the study to detect a mean difference of 10 mg of morphine between the two groups

Secondary outcome measures include: Pain evaluation with the use of VAS at rest, VAS on walking and on knee flexion; functional outcome evaluation with the 6 min walk tests, degree of knee flexion, Scores obtained in self-assessment questionaire (WOMAC-Western Ontario and McMaster University questionaire for knee osteoarthritis and CHAMPS-Community Healthy Activities Model Program for Seniors). These values will be compared with baseline values recorded before surgery.

It is hypothesized that PRF and TRF of the saphenous nerve and genicular nerves to the knee joint can improve the early and late functional recovery and the pain control after TKA when compared with the CACB

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of knee Osteoarthritis requiring Total Knee Arthroplasty (TKA)

Exclusion Criteria:

* Previous TKA (revision surgery)
* ASA (American Society of Anesthesiology) Classification > 3
* Known Rheumatologic disease
* Morbid Obesity (BMI > 45)
* Inability to perform simple physical tasks (6 minutes walk test, Timed-Up and Go test)
* Organ transplant, Allergy to opioids, to local anesthetics or other medications used in the study,
* Chronic use of opioids or sedatives, Contraindication to receive regional anesthesia (e.g. coagulation defect), contraindication to Patient Controlled Analgesia pump (PCA) or inability to use PCA or to comprehend pain scales

Ages: 45 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2015-09-14 (Actual); Primary Completion 2017-06-02 (Actual); Study Completion 2017-07-07 (Actual)

PRIMARY OUTCOMES:
Postoperative morphine consumption | first postoperative day (first 24 hours)

SECONDARY OUTCOMES:
Timed-Up and Go Test | 2nd postoperative day
  TUG measures the time that a person takes to rise from a chair, walk three meters, turn around, walk back to the chair, and sit down. During the test, the person is expected to use any mobility aids that they would normally require
Six minutes walk test | 6 weeks after surgery
  This test measures the distance that a patient can quickly walk on a flat, hard surface in a period of 6 minutes
Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC) | 6 weeks after surgery
  The WOMAC consists of 24 items divided into 3 subscales: Pain (5 items);Stiffness (2 items); Physical Function (17 items).
  The Extent of pain, stiffness in the knee, and physical function related to the disability due to the knee osteoarthritis are assessed with the WOMAC index, before and 6 weeks after surgery (Western-Ontario-McMaster-Universities-Osteoarthritis-Index).
Visual Analogue Scale (VAS) for pain at rest | 6 weeks after surgery
Visual Analogue Scale (VAS) for pain at movement | 6 weeks after surgery
Pain medication consumption | 6 weeks after surgery
Visual Analogue Scale (VAS) for pain at rest | first 24 hours after surgery
Visual Analogue Scale (VAS) for pain at movement | First 24 hours after surgery
CHAMPS (Community Healthy Activities Model Program for Seniors) questionnaire | 6 weeks after surgery

CONTACTS AND LOCATIONS:
Overall Officials: Francesco Carli, Professor, Study Director — Mc Gill Univeristy Health Center; Juan Francisco Asenjo, Professor, Principal Investigator — Mc Gill Univeristy Health Center
Locations (1):
- McGill University Health Centre, Montreal General Hospital, Montreal, Quebec, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Patterson ME, Bland KS, Thomas LC, Elliott CE, Soberon JR Jr, Nossaman BD, Osteen K. The adductor canal block provides effective analgesia similar to a femoral nerve block in patients undergoing total knee arthroplasty--a retrospective study. J Clin Anesth. 2015 Feb;27(1):39-44. doi: 10.1016/j.jclinane.2014.08.005. Epub 2014 Nov 22. PMID 25468584
- [Result] Machi AT, Sztain JF, Kormylo NJ, Madison SJ, Abramson WB, Monahan AM, Khatibi B, Ball ST, Gonzales FB, Sessler DI, Mascha EJ, You J, Nakanote KA, Ilfeld BM. Discharge Readiness after Tricompartment Knee Arthroplasty: Adductor Canal versus Femoral Continuous Nerve Blocks-A Dual-center, Randomized Trial. Anesthesiology. 2015 Aug;123(2):444-56. doi: 10.1097/ALN.0000000000000741. PMID 26079800
- [Result] Carli F, Clemente A, Asenjo JF, Kim DJ, Mistraletti G, Gomarasca M, Morabito A, Tanzer M. Analgesia and functional outcome after total knee arthroplasty: periarticular infiltration vs continuous femoral nerve block. Br J Anaesth. 2010 Aug;105(2):185-95. doi: 10.1093/bja/aeq112. Epub 2010 Jun 14. PMID 20551021
- [Result] Shah NA, Jain NP. Is continuous adductor canal block better than continuous femoral nerve block after total knee arthroplasty? Effect on ambulation ability, early functional recovery and pain control: a randomized controlled trial. J Arthroplasty. 2014 Nov;29(11):2224-9. doi: 10.1016/j.arth.2014.06.010. Epub 2014 Jun 19. PMID 25041873
- [Result] Jaeger P, Zaric D, Fomsgaard JS, Hilsted KL, Bjerregaard J, Gyrn J, Mathiesen O, Larsen TK, Dahl JB. Adductor canal block versus femoral nerve block for analgesia after total knee arthroplasty: a randomized, double-blind study. Reg Anesth Pain Med. 2013 Nov-Dec;38(6):526-32. doi: 10.1097/AAP.0000000000000015. PMID 24121608